CLINICAL TRIAL: NCT03495076
Title: Perceptual Distortions in Acute Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Collaborators: University of Luebeck (Other)
Responsible Party: Principal Investigator, Wacław Adamczyk, Principal Investigator, main director of the project, The Jerzy Kukuczka Academy of Physical Education in Katowice
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 1/2018
Record Dates: First submitted 2018-03-28; First posted 2018-04-11 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Neck Pain, Posterior; Pain, Acute
Keywords: Tactile acuity; Tactile dysfunction; Sensory dissociation; Two-point discrimination; Perception
MeSH Terms: conditions — Neck Pain; Acute Pain | interventions — Sodium Chloride; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Within-group designed study. All participants will be assessed in three different experimental conditions (control, saline injection, sham injection). The order of conditions will be counterbalanced across participants and randomly chosen.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be informed about the hypotheses tested and will not be informed about the sham-injection condition. The fact that they received only one injection during the study period will be uncovered at the end of the project.
  Examiner will be blinded towards conditions sequence. Between pre-test and post-test examiner will not be present in the research room to provide blinding towards the manipulation provided (control, saline injection, sham injection).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Saline injection (Experimental): In the saline condition, acute neck pain will be induced via 0.5 ml hypertonic (5% NaCl) saline solution.
  Interventions: Other: Saline injection
- Sham injection (Sham Comparator): In the sham injection condition, a real needle will be shown to the participants to imitate and produce the anticipation of a pain experience.
  Interventions: Other: Sham injection
- Control (No Intervention): Participants in the control condition will not receive any kind of pain or pinprick sensation.

INTERVENTIONS:
Other: Saline injection — In the saline injection condition, acute neck pain will be induced via 0.5 ml hypertonic (5% NaCl) saline bolus injection which is a commonly used model of acute pain. Saline will be injected into the right (or left) trapezius muscle at the level of C7 cervical level. Injections will be performed by a physician under ultrasound imaging guidance to ensure that each single injection will be equally placed at the same depth. The side for the pain induction will be randomised across subjects. The place of needle insertion and corresponding point on the opposite side of the body will be covered by placing a small piece of adhesive plaster to ensure blinding.
  Other Names: Pain induced by saline injection
  Arms: Saline injection
Other: Sham injection — In the sham-injection condition (nocebo comparator), a real needle will be shown to the participants to imitate and produce the anticipation of a pain experience. A pinprick sensation will be produced by a weighted stimulus applied perpendicularly to the skin without piercing the skin. A stimulus of 512 millinewtons (mN) will be used to produce a pinprick sensation and activation of cutaneous nociceptors. Adhesive tapes covering stimulation points will also be provided. The stimuli will be applied in exactly the same spot as the real injection in previous experimental condition.
  Other Names: Pain induced by sham injection
  Arms: Sham injection

SUMMARY:
Research has shown that chronic pain is related to variety of perceptual distortions. Little is known on how acute pain experience influences perception, especially precision of touch. This project is aiming to test the hypothesis of pain as a process of biological value leading to improvement in tactile acuity.

DETAILED DESCRIPTION:
This project has following goals:

1. To test the hypothesis of pain as a process of biological value leading to improvement in tactile acuity
2. To investigate intra-rater reliability of tests measuring perceptual distortions in pain
3. To investigate validity of novel tests measuring perceptual distortions in pain
4. To explore the influence of acute neck pain on left/right recognition task
5. To explore the effect of acute neck pain on body perception

ELIGIBILITY:
Inclusion Criteria:

* Only participants without tactile dysfunction will be included.
* Participants reporting availability during the days in which the research will be performed.

Exclusion Criteria:

* current pain experience
* episodes of neck
* thoracic or lumbar pain lasting more than 24 hours within previous month
* history of chronic pain, i.e. pain lasting more than three-month period
* comorbidities affecting nervous system
* cardio-vascular diseases
* psychiatric illnesses
* any disease requiring systematic drug consumption
* diagnosed scoliosis.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Tactile acuity measured by two-point discrimination test (TPD). | TPD change from baseline at 30 seconds post-manipulation period (e.g. saline injection).
  Mechanical callipers will be delicately applied to the spot just below the location where real or sham injection will be administered. Tactile stimuli will be applied until the very first blanching of the skin. Testing will be commenced with 0 mm between the two calliper's tips, and then the distance between them will be gradually increased until participants will able to verbally report that two points had been touched instead of one. Subsequently, the descending sequence will be applied until the perception of the two points disappeared.

SECONDARY OUTCOMES:
Laterality judgements measured by left/right recognition application. | Measured at baseline and ~30 seconds after manipulation (e.g. saline injection).
  A set of images displaying human neck in different orientation in space will be show to participants. The goal of the task is to decide whether given picture depicts neck rotated to the left or right or flexed into left o right side. The accuracy and response time is measured.
Sensory dissociation measured by two-point estimation task (TPE). | Measured at baseline and ~30 seconds after manipulation (e.g. saline injection).
  One tactile stimulus will be applied until the very first blanching of the skin, with a 120 mm horizontal separation between the calipers' tips. Participants will be then asked to indicate with their calipers the distance they have perceived.

OTHER OUTCOMES:
Pain intensity measured behaviourally on a Numerical Rating Scale (NRS). | Pain intensity will be measured just after saline/sham injection and every 10 seconds after this time point up until 30 seconds.
  The scale for pain intensity ratings will range from 0 = "no pain" to 10 = "the worst pain imaginable"
Distribution of pain measured by estimating the diameter of the circle representing area affected by pain. | Pain distribution will be measured just after saline/sham injection and every 10 seconds after this time point up until 30 seconds.
  Greater circle (diameter in cm) will refer to the greater distribution of pain (larger body surface affected).
Fear of pain measured on a Numerical Rating Scale (NRS) | Fear of pain (state) measured only at baseline
  Fear of pain will be rated on a scale ranging from 0 = "not at all" to 10 = "very much".
Fear of Pain Questionnaire (FPQ-III). | Measured only at baseline.
  FPQ-III consists of three subscales measuring: minor pain, severe pain, and medical pain. Each subscale contains 10 items. The total score has a range 30-150. A higher score indicates greater fear of pain.
Pain duration | One measurement collected immediately after pain alleviation. The time frame will vary from person to person, however it is expected to collect the data an average 10 minutes after the injection.
  Pain duration measured by physician in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Wacław M Adamczyk, MSc, Study Director — The Jerzy Kukuczka Academy of Physical Education, Department of Physiotherapy
Locations (1):
- The Jerzy Kukuczka Academy of Physical Education, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adamczyk WM, Saulicz O, Saulicz E, Luedtke K. Tactile acuity (dys)function in acute nociceptive low back pain: a double-blind experiment. Pain. 2018 Mar;159(3):427-436. doi: 10.1097/j.pain.0000000000001110. PMID 29140929
- [Background] Adamczyk WM, Luedtke K, Saulicz O, Saulicz E. Sensory dissociation in chronic low back pain: Two case reports. Physiother Theory Pract. 2018 Aug;34(8):643-651. doi: 10.1080/09593985.2017.1423431. Epub 2018 Jan 11. PMID 29324082
- [Background] Adamczyk W, Luedtke K, Saulicz E. Lumbar Tactile Acuity in Patients With Low Back Pain and Healthy Controls: Systematic Review and Meta-Analysis. Clin J Pain. 2018 Jan;34(1):82-94. doi: 10.1097/AJP.0000000000000499. PMID 28328700
- [Background] Harvie DS, Edmond-Hank G, Smith AD. Tactile acuity is reduced in people with chronic neck pain. Musculoskelet Sci Pract. 2018 Feb;33:61-66. doi: 10.1016/j.msksp.2017.11.009. Epub 2017 Nov 21. PMID 29180111
- [Background] Elsig S, Luomajoki H, Sattelmayer M, Taeymans J, Tal-Akabi A, Hilfiker R. Sensorimotor tests, such as movement control and laterality judgment accuracy, in persons with recurrent neck pain and controls. A case-control study. Man Ther. 2014 Dec;19(6):555-61. doi: 10.1016/j.math.2014.05.014. Epub 2014 Jun 10. PMID 24957711